CLINICAL TRIAL: NCT07015632
Title: Quantitative Analysis of Upper Extremity Functional Movement of the Upper Extremity in Patients With Duchenne Muscular Dystrophy
Brief Title: ML-Based Multi-Sensor Fall Risk Screening in DMD
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Hyung Lee, Clinical Assistant Professor, Seoul National University Hospital
Other Study IDs: 0420232060
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: DMD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Performance of the Upper Limb, Brooke Scale, grip strength test — Thirty patients will be evaluated at three time points (baseline, 6 months, 12 months) using clinical assessments (PUL 2.0, Brooke Scale, grip strength), computer vision-based video analysis, and machine learning algorithms.

SUMMARY:
This prospective observational study aims to analyze changes in upper extremity functional movement over time in children with Duchenne Muscular Dystrophy (DMD). Thirty patients will be evaluated at three time points (baseline, 6 months, 12 months) using clinical assessments (PUL 2.0, Brooke Scale, grip strength), computer vision-based video analysis, and machine learning algorithms. The goal is to improve future upper limb evaluation methods for non-ambulatory DMD patients. The study includes safety monitoring and adheres to ethical standards, ensuring patient data confidentiality and providing compensation if adverse effects occur.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a confirmed genetic diagnosis of Duchenne Muscular Dystrophy (DMD)
2. Age over 10 and under 30 years
3. Brooke Scale score between 2 and 5
4. Manual muscle test grade below 3 for shoulder abduction muscles

Exclusion Criteria:

1. Individuals who are unable or unwilling to provide informed consent
2. Brooke Scale score of 1 or 6
3. Individuals with cognitive impairments that significantly limit their ability to participate in assessments

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: South Korea
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Performance of the upper limb module 2.0 | baseline - 6 months - 12 months
  The Performance of the Upper Limb (PUL) Module 2.0 is a validated assessment tool designed to evaluate upper limb function in individuals with Duchenne Muscular Dystrophy. The PUL 2.0 consists of 22 items covering three domains: shoulder level, mid-level (elbow), and distal level (hand). Each item is scored based on task performance, and the total score ranges from 0 to 42, with higher scores indicating better upper limb function.

SECONDARY OUTCOMES:
Brooke score | baseline - 6 months - 12 months
  The Brooke Upper Extremity Functional Rating Scale is a 6-point scale used to evaluate upper limb functional ability, primarily in patients with neuromuscular disorders such as Duchenne Muscular Dystrophy. Scores range from 1 to 6, where:
  1 = Able to abduct arms in a full circle until they touch above the head 6 = Cannot raise hands to the mouth and has no useful function of the hands
  Lower scores indicate better upper limb function.
grip strength | baseline - 6 months - 12 months
  Grip strength will be measured using the Jamar Plus+ Digital Hand Dynamometer, a validated and widely used device for quantifying hand grip strength in kilograms (kg). Participants will be instructed to sit upright with the shoulder adducted and neutrally rotated, elbow flexed at 90 degrees, forearm in neutral position, and wrist in 0 to 30 degrees extension. The average of three consecutive trials will be recorded for each assessment. Higher values indicate greater grip strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno, South Korea

IPD SHARING:
Plan to Share IPD: No